CLINICAL TRIAL: NCT00705341
Title: MethaCholine Bronchoprovocation - Influence of High Potency Inhaled corticoSteroids in Asthma (MeCIS) Study
Brief Title: MethaCholine Bronchoprovocation Study (MeCIS)
Acronym: MeCIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Washington University School of Medicine (Other); St. Louis University (Other); Long Island Jewish Medical Center (Other); North Shore University Hospital (Other); Baylor College of Medicine (Other); University of Vermont (Other); Nemours Children's Clinic (Other); University of Florida (Other); Indiana University (Other); Ohio State University (Other); NYU Langone Health (Other); University of Missouri-Columbia (Other); Northwestern University (Other); Louisiana State University Health Sciences Center in New Orleans (Other); University of Miami (Other); University of South Florida (Other); University of California, San Diego (Other); National Jewish Health (Other); Duke University (Other)
Responsible Party: Principal Investigator, Janet Holbrook, Associate Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: ALAACRC07
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Asthma
Keywords: Normal Controls
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose fluticasone for phase 2 (Active Comparator): For people with asthma, fluticasone at 250 mcg per day; phase 2 of study
  Interventions: Drug: fluticasone
- High dose fluticasone for phase 2 (Active Comparator): For people with asthma, fluticasone at 1000 mcg per day; phase 2 of study
  Interventions: Drug: fluticasone
- Nonasthmatic controls for phase 1 (No Intervention): People without asthma will be enrolled to perform 1 methacholine challenge test in phase 1 of the study
- Asthmatic controls for phase 1 (No Intervention): People with asthma will be enrolled to perform 1 methacholine challenge test in phase 1 of the study

INTERVENTIONS:
Drug: fluticasone — Inhaled corticosteroid approved for treatment of asthma
  Other Names: Flovent diskus
  Arms: High dose fluticasone for phase 2; Low dose fluticasone for phase 2

SUMMARY:
The purpose of this research is to evaluate the methacholine challenge test as an accurate indicator of asthma in patients receiving treatment for asthma. Phase 1 on the study compares methacholine challenge test results from asthma patients to those from people who do not have asthma. In phase 2, test results for people with asthma on low dose inhaled corticosteroid will be compared to results on high dose inhaled corticosteroids. Both males and females with stable asthma (asthma participants) and without asthma (controls) enrolled. Participants will be between 12 and 69 years of age.

DETAILED DESCRIPTION:
The study consists of two phases. The first phase is a cross-sectional, case-control study measuring the sensitivity and specificity of methacholine challenge testing for differentiating asthmatic participants from non-asthmatic controls. The second phase is a cross-over, randomized, double-masked trial designed to evaluate the impact of high dose versus low dose inhaled corticosteroids (ICS) on bronchial hyperreactivity (BHR) in asthmatics.

ELIGIBILITY:
Asthmatic participants

Inclusion Criteria:

* Males or females greater than or equal to 12 and less than 70 years of age
* Physician-diagnosed and investigator-confirmed stable asthma (excluding exercise induced asthma)
* Current treatment for asthma by a healthcare provider within the preceding twelve months: current asthma treatment defined as regular use of asthma medications. Asthma medications include short and long acting adrenergic bronchodilators, bronchodilator combinations, inhaled anticholinergics, inhaled corticosteroids, cromolyn sodium and nedocromil, leukotriene modifiers and methylxanthines
* Stable asthma defined by no asthma exacerbation (emergency room visit, hospitalization, course of increased systemic steroids, or urgent health care visit for asthma) during the prior four weeks
* Forced expiratory volume at one second (FEV1) >70% predicted pre-bronchodilator
* Ability to provide screening and baseline information
* Ability and willingness to provide informed consent
* For women of childbearing potential: not pregnant, non-lactating, and agree to practice an adequate birth control method (abstinence, combination barrier and spermicide, or hormonal) for the duration of the study

Exclusion Criteria:

* Chronic oral steroid therapy (daily)
* Oral corticosteroid use within past 4 weeks
* Respiratory tract infection within past 4 weeks
* Chronic diseases (other than asthma) that in the opinion of the investigator would prevent participation in the trial or put the participant at risk by participation, e.g. chronic diseases of the lung (other than asthma), heart, liver, kidney, or nervous system, or immunodeficiency
* Known allergy to methacholine (for example, a previous bad reaction to methacholine) or to any other parasympathomimetic agents
* Current use of beta adrenergic blocking agent (a heart medicine) or a cholinesterase inhibitor (medicine used to treat myasthenia gravis or Alzheimer's disease).
* History of epilepsy, cardiovascular disease with bradycardia (slow heart beat), vagotonia (increased activity of the vagus nerve causing slow heart rate or low blood pressure), peptic ulcer disease, thyroid disease, or urinary tract obstruction
* History of cigarette smoking within the past 5 years or >10 pack years total
* Use of investigative drugs or intervention trials in the 30 days prior to enrollment or during the duration of the study
* Any condition or compliance issue which in the opinion of the investigator might interfere with participation

Nonasthmatic control criteria:

Inclusion Criteria:

* Males or females greater than or equal to 12 and less than 70 years of age
* Individuals who are in good overall health
* Age (within ten years for above 25 years of age and +/- five years for 12-25 years of age) and sex matched to the asthmatic group

Exclusion Criteria:

* A subject will be excluded if there is a history within the previous 5 years of:

  * clinically diagnosed allergy (allergic rhinitis, hay fever or atopic dermatitis),
  * asthma (beyond 6 years of age),
  * chronic nasal or sinus disease, or
  * other chronic lung diseases
* Respiratory tract infection within past 4 weeks
* History of cigarette smoking within the past 5 years or >10 pack years total
* Known allergy to methacholine (for example, a previous bad reaction to methacholine) or to any other parasympathomimetic agents
* Current use of beta adrenergic blocking agent (a heart medicine) or a cholinesterase inhibitor (medicine used to treat myasthenia gravis or Alzheimer's disease).
* History of epilepsy, cardiovascular disease with bradycardia (slow heart beat), vagotonia (increased activity of the vagus nerve causing slow heart rate or low blood pressure), peptic ulcer disease, thyroid disease, or urinary tract obstruction

Ages: 12 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaharu Sumino, MD, Principal Investigator — St. Louis Asthma Clinical Research Center
Locations (13):
- United States (13):
  - University of California at San Diego, San Diego, California
  - The Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami/Univestiy of South Florida, Miami, Florida
  - Northwestern University Memorial Hospital, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Louisianna State University, New Orleans, Louisiana
  - University of Missouri-Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Consortium/Columbia University, New York, New York
  - New York Medical College, Valhalla, New York
  - Ohio State University, Columbus, Ohio
  - Vermont Lung Center at the University of Vermont, Burlington, Vermont

REFERENCES:
- [Derived] Sumino K, Sugar EA, Irvin CG, Kaminsky DA, Shade D, Wei CY, Holbrook JT, Wise RA, Castro M; American Lung Association Asthma Clinical Research Centers. Methacholine challenge test: diagnostic characteristics in asthmatic patients receiving controller medications. J Allergy Clin Immunol. 2012 Jul;130(1):69-75.e6. doi: 10.1016/j.jaci.2012.02.025. Epub 2012 Apr 1. PMID 22465214
- See also: Asthma Clinical Research Centers website — http://cctrials.org/alaacrc

RESULTS

PARTICIPANT FLOW:
Groups:
- Asthmatic Controls for Phase 1: People with asthma perform 1 methacholine challenge test in phase 1 to measure the sensitivity and specificity of methacholine challenge testing. Participants did not receive an intervention in phase 1.
- Non Asthmatic Controls for Phase 1: People without asthma perform 1 methacholine challenge test in phase 1 to measure the sensitivity and specificity of methacholine challenge testing. Participants did not receive an intervention in phase 1.
- Low Dose, Then High Dose Fluticasone for Phase 2: People with asthma receive fluticasone at 250 mcg per day (28 days), then wash-out period (28 days), then fluticasone at 1000 mcg per day (28 days) in phase 2.
- High Dose, Then Low Dose Fluticasone for Phase 2: People with asthma receive fluticasone at 1000 mcg per day 28 days), then wash-out period (28 days), fluticasone at 250 mcg per day (28 days) in phase 2.
Period: Phase 1:Control Challenge
Arm/Group | Asthmatic Controls for Phase 1 | Non Asthmatic Controls for Phase 1 | Low Dose, Then High Dose Fluticasone for Phase 2 | High Dose, Then Low Dose Fluticasone for Phase 2
Started | 126 | 93 | 0 | 0
Completed | 126 (If participants in this group met criteria, they were randomized into phase 2) | 93 (Nonasthmatic controls did not advance to phase 2 due to design of study) | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase 2: Trial
Arm/Group | Asthmatic Controls for Phase 1 | Non Asthmatic Controls for Phase 1 | Low Dose, Then High Dose Fluticasone for Phase 2 | High Dose, Then Low Dose Fluticasone for Phase 2
Started | 0 | 0 | 30 (This group was randomized from asthmatic controls in phase 1 if they met criteria to be in phase 2) | 32 (This group was randomized from asthmatic controls in phase 1 if they met criteria to be in phase 2)
Completed | 0 | 0 | 23 | 28
Not Completed | 0 | 0 | 7 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 4
Not completed — Did not meet post-diluent threshold | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nonasthmatic Controls for Phase 1: People without asthma perform 1 methacholine challenge test in phase 1 to measure the sensitivity and specificity of methacholine challenge testing. Participants did not receive an intervention in phase 1.
- Total: Total of all reporting groups
Arm/Group | Nonasthmatic Controls for Phase 1 | Asthmatic Controls for Phase 1 | Total
Number analyzed (Participants) | 93 | 126 | 219
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 93 | 126 | 219
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33 (13) | 38 (15) | 35 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 84 | 140
  Male | 37 | 42 | 79
Region of Enrollment [Number; unit: participants]
  United States | 93 | 126 | 219

OUTCOME MEASURES:

1. Primary Outcome: Methacholine Challenge Test Result for Phase 2
Description: Presence and degree of airway hyperresponsiveness assessed by methacholine challenge test post-diluent baseline (PC20) after medication holds; PC20 is the methacholine dose at which the amount of air expired in the first second during a forced expiratory maneuver is reduced by 20%; value represents change in baseline to 4 weeks
Time Frame: weeks 0, 4
Population: There was a significant period effect in the percentage change in post diluent baseline (PC20) for high- and low-dose depending upon the order in which the doses were administered. In order to remove the effect of the order, we compared the high- and low-dose MCT results exclusively during the first cross over.
Measure: Geometric Mean (Full Range); unit: mg/ml
Groups:
- 4 Weeks of High Dose Fluticasone: 4 weeks of Fluticasone (Flovent diskus) 500 mcg twice daily (1000mcg/day)
- 4 Weeks of Low Dose Fluticasone: 4 weeks of Fluticasone (Flovent diskus) 250 mcg once daily
Arm/Group | 4 Weeks of High Dose Fluticasone | 4 Weeks of Low Dose Fluticasone
Number analyzed (Participants) | 28 | 23
mg/ml | 1.19 [0.10 to 26.92] | 2.04 [0.16 to 48.00]
Statistical Analysis 1: Comparison: 4 Weeks of High Dose Fluticasone vs 4 Weeks of Low Dose Fluticasone; Log-linear generalized estimating equation (GEE) models were used to assess the dose effect on PC20; Test type: Superiority or Other; p = 0.65, Regression, Linear

2. Secondary Outcome: Predictive Value of Methacholine Challenge Test for Phase 1
Description: Predictive value of methacholine challenge test in phase 1 for asthmatics and nonasthmatic controls
Time Frame: one time
Measure: Number (95% Confidence Interval); unit: % predictive value
Arm/Group | Asthmatic Controls for Phase 1 | Non Asthmatic Controls for Phase 1
Number analyzed (Participants) | 126 | 93
% predictive value | 96 [90 to 99] | 75 [66 to 83]

ADVERSE EVENTS:
Description: Adverse events were not collected in phase 1 of the study
Groups:
- Low Dose for phase1: 4 weeks of Fluticasone (Flovent diskus) 250 mcg twice daily (500 mcg/day)
- High Dose for Phase 2: 4 weeks of Fluticasone (Flovent diskus) 500 mcg twice daily (1000mcg/day)
Arm/Group | Low Dose for phase1 | High Dose for Phase 2
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 23/30 | 22/32
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose for phase1 (N=30) | High Dose for Phase 2 (N=32)
headache (General disorders) | 22 | 22
Oral candidiasis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 23 | 22
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 18 | 19
Sinusitis (Infections and infestations) | 5 | 4
Pharyngitis (General disorders) | 13 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 19
Hoarseness/ dysphoria (General disorders) | 12 | 16
Upper respiratory infection (Infections and infestations) | 7 | 6
Upper respiratory inflammation (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Viral lower respiratory infection (Infections and infestations) | 2 | 5
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Gastrointestinal discomfort and pain (Gastrointestinal disorders) | 10 | 9
Viral gastrointestinal infection (Infections and infestations) | 1 | 1
Nausea and vomiting (Gastrointestinal disorders) | 8 | 5
Diarrhea (Gastrointestinal disorders) | 4 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 10
Muscle injury (Musculoskeletal and connective tissue disorders) | 3 | 6
Influenza (Infections and infestations) | 2 | 4
Fever (Infections and infestations) | 6 | 6
Injury (Injury, poisoning and procedural complications) | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No